CLINICAL TRIAL: NCT04365634
Title: A Single-center Retrospective Study to Find Prediction Factors Related to Mortality of COVID-19 Patients by Univariate and Multivariate Analysis.
Brief Title: A Single-center Retrospective Study to Find Prediction Factors Related to Mortality of COVID-19 Patients.
Status: Completed | Type: Observational
Sponsor: Tongji Hospital (Other)
Responsible Party: Principal Investigator, Qin Ning, Professor, Tongji Hospital
Other Study IDs: TJ20200202
Record Dates: First submitted 2020-04-25; First posted 2020-04-28 (Actual); Last update posted 2020-04-28 (Actual); Status verified 2020-04

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Diabetes: Diabetes mellitus was diagnosed according to the standards of American Diabetes Association which were briefly described as FPG ≥ 7.0 mmol/L (Fasting is defined as no caloric intake for at least 8 h) or 2-h plasma glucose ≥ 11.1 mmol/L during Oral glucose tolerance test (OGTT), or with classic symptoms of hyperglycemia or hyperglycemic crisis, a random plasma glucose (RPG) ≥ 11.1 mmol/L. And in this group, we have 129 COVID-19 patients with diabetes.
- Non-diabetes: Patients who do not meet the American Diabetes Association's standard diagnosis of diabetes are defined as non-diabetes. And in this group, we have 177 COVID-19 patients without diabetes.
- Survivors: COVID-19 patients who survived on the 28th day in hospital belong to survivors group. In the survivors group, we included 201 patients with complete data.
- Non-survivors: COVID-19 patients who did not survive on the 28th day in hospital belong to non-survivors group. In the non-survivors group, we included 54 patients with complete data.

SUMMARY:
In the single-centered, retrospective study, 306 hospital patients (including 129 diabetes and 177 non-diabetes patients) confirmed with SARS-CoV-2 infection were enrolled in Tongji Hospital, Wuhan, China. Clinical characteristics including clinical manifestation, laboratory parameters, lung CT features and clinical outcomes were compared between diabetes and non-diabetes patients. The prediction factors were analyzed for mortality of COVID-19 by univariate and multivariate analysis.

ELIGIBILITY:
Inclusion Criteria:

Patients admitted from Feb 2, 2020 to Feb 15, 2020, diagnosed with SARS-CoV-2 pneumonia according to interim guidance of National health commission of the people's republic of China.

Exclusion Criteria:

With SARS-CoV-2 RNA detection negative results.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The patients admitted from Feb 2, 2020 to Feb 15, 2020, diagnosed with SARS-CoV-2 pneumonia according to interim guidance of National health commission of the people's republic of China were enrolled. Laboratory confirmed cases were identified with positive viral RNA by real-time RT-PCR detection by the local health authority or our hospital from specimen taken from throat or nasal swab.
Sampling Method: Probability Sample
Enrollment: 306 (Actual)
Dates: Start 2020-02-02 (Actual); Primary Completion 2020-03-15 (Actual); Study Completion 2020-04-01 (Actual)

PRIMARY OUTCOMES:
Find the prediction factors associated with hospitalized death of patients with COVID-19 by univariate and multivariate analysis | 28 days

SECONDARY OUTCOMES:
Demographics and clinical characteristics | 28 days
Laboratory parameters and radiography image features | 28 days
Treatment, complications and clinical outcomes | 28 days

CONTACTS AND LOCATIONS:
Overall Officials: Meifang Han, Professor, Study Chair — Tongji Hospital
Locations (1):
- Tongji Hospital, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Han M, Ma K, Wang X, Yan W, Wang H, You J, Wang Q, Chen H, Guo W, Chen T, Ning Q, Luo X. Immunological Characteristics in Type 2 Diabetes Mellitus Among COVID-19 Patients. Front Endocrinol (Lausanne). 2021 Mar 11;12:596518. doi: 10.3389/fendo.2021.596518. eCollection 2021. PMID 33776910